CLINICAL TRIAL: NCT03971474
Title: A Phase II Randomized Study of Ramucirumab Plus MK3475 (Pembrolizumab) Versus Standard of Care for Patients Previously Treated With Immunotherapy for Stage IV or Recurrent Non-Small Cell Lung Cancer (Lung-MAP Non-Matched Sub-Study)
Brief Title: Ramucirumab and Pembrolizumab Versus Standard of Care in Treating Patients With Stage IV or Recurrent Non-small Cell Lung Cancer (A Lung-MAP Non-Match Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1800A; NCI-2019-00703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1800A (Other: SWOG); S1800A (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; Gemcitabine; pembrolizumab; Pemetrexed; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed) (Active Comparator): Patients receive docetaxel IV over 10-30 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 or ramucirumab IV over 60 minutes and docetaxel IV over 10-30 minutes on day 1. Patients with non-squamous NSCLC receiving docetaxel and gemcitabine hydrochloride, also receive pemetrexed IV over 10 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Drug: Pemetrexed; Drug: Pemetrexed Disodium; Biological: Ramucirumab
- Arm B (ramucirumab, pembrolizumab) (Experimental): Patients receive ramucirumab IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Biological: Ramucirumab

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
  Arms: Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm B (ramucirumab, pembrolizumab)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate
  Arms: Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed)
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
  Arms: Arm A (docetaxel, gemcitabine, ramucirumab, pemetrexed)
Biological: Ramucirumab — Given IV
  Other Names: anti-VEGFR-2 fully human monoclonal antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase II Lung-MAP non-Match treatment trial studies how well ramucirumab and pembrolizumab work versus standard of care in treating patients with non-small cell lung cancer that is stage IV or has come back. Immunotherapy with monoclonal antibodies, such as ramucirumab and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in standard of care chemotherapy for non-small cell lung cancer, such as docetaxel, gemcitabine hydrochloride, and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ramucirumab and pembrolizumab together may work better in treating patients with non-small lung cancer compared to standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival between patients previously treated with platinum-based chemotherapy and immunotherapy for stage IV or recurrent non-small cell lung cancer randomized to ramucirumab and MK-3475 (pembrolizumab) versus standard of care (SoC).

SECONDARY OBJECTIVES:

I. To compare response rates between the arms, including complete response (CR) and partial response (PR) (confirmed and unconfirmed).

II. To compare the disease control rate (CR, PR, confirmed and unconfirmed and stable disease [SD]).

III. To evaluate the duration of response (DoR) among responders within each arm.

IV. To evaluate the frequency and severity of toxicities within each arm. V. To compare investigator assessed-progression-free survival (IA-PFS) between the arms.

VI. To evaluate the clinical outcomes (overall survival [OS], IA-PFS, response) by randomization stratification factors by comparing outcomes within the ramucirumab and MK-3475 (pembrolizumab) arm, performing a sub-group analysis of the arms, and by evaluating an interaction between the factors and treatment arm.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate if PD-L1 expression levels are associated with clinical outcomes (OS, IA-PFS, and response).

II. To evaluate if tumor mutation burden (TMB) as determined by the Foundation Medicine Inc (FMI) Foundation One panel is associated with clinical outcomes.

III. To collect, process, and bank cell-free (circulating cell-free deoxyribonucleic acid [cfDNA]) at baseline and progression for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor DNA (ctDNA).

IV. To establish a tissue/blood repository to pursue future studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients may receive docetaxel intravenously (IV) over 10-30 minutes on day 1, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, pemetrexed IV over 10 minutes on day 1 (non-squamous NSCLC patients only), or ramucirumab IV over 60 minutes combined with docetaxel IV over 10-30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive ramucirumab IV over 60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment (prior to disease progression), patients are followed up every 3 months for the first year, and then every 6 months for up to 3 years from date of randomization. After completion of study treatment (after disease progression), patients are followed up every 6 months for 2 years, then at the end of year 3 from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been assigned to S1800A by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Patients who were screened under S1400 (legacy screening/pre-screening study) must have had prior PD-L1 testing by the Dako 22C3 PharmDx immunohistochemistry (IHC) assay, and must have results available for stratification purposes
* Patients must not have EGFR sensitizing mutations, EGFR T790M mutation, ALK gene fusion, ROS 1 gene rearrangement, and BRAF V600E mutation unless they have progressed following all standard of care targeted therapy
* Patients must not have an active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patients must not have any history of primary immunodeficiency
* Patients must not have experienced the following:

  * Any grade 3 or worse immune-related adverse event (irAE). Exception: asymptomatic nonbullous/nonexfoliative rash
  * Any unresolved grade 2 irAE
  * Any toxicity that led to permanent discontinuation of prior anti-PD-1/PD-L1 immunotherapy

    * Exception to the above: Toxicities of any grade that requires replacement therapy and has stabilized on therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are allowed
* Patients must not have any history of organ transplant that requires use of immunosuppressives
* Patients must not have clinical signs or symptoms of active tuberculosis infection
* Patients must not have history of (non-infectious) pneumonitis that required steroids or current pneumonitis/interstitial lung disease
* Patients must not have had a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to sub-study randomization
* Patients must not have a history of gastrointestinal perforation or fistula within six months prior to sub-study randomization
* Patients must not have grade 3-4 gastrointestinal bleeding (defined by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5) within three months prior to sub-study randomization
* Patients must not have any known allergy or reaction to any component of the investigational and standard of care formulations
* Patients must not have any grade III/IV cardiac disease as defined by the New York Heart Association criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within six months prior to sub-study randomization, or serious uncontrolled cardiac arrhythmia
* Patients must not have experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within six months prior to sub-study randomization
* Patients must not have documented evidence of acute hepatitis or have an active or uncontrolled infection
* Patients with known human immunodeficiency virus (HIV) infection are eligible, provided they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to randomization
* Patients with evidence of chronic hepatitis B virus (HBV) infection are eligible provided viral load is undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients must not have undergone major surgery within 28 days prior to sub-study randomization, or subcutaneous venous access device placement within 7 days prior to randomization. Any patient with postoperative bleeding complications or wound complications from a surgical procedure performed in the last two months should be excluded. The patient must not have elective or planned major surgery to be performed during the course of the clinical trial
* Patients must not have gross hemoptysis within two months of sub-study randomization (defined as bright red blood or >= 1/2 teaspoon) or with radiographic evidence of intratumor cavitation or has radiologically documented evidence of major blood vessel invasion or encasement by cancer
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must not have been diagnosed with venous thrombosis less than 3 months prior to randomization. Patients with venous thrombosis diagnosed more than 3 months prior to randomization must be on stable doses of anticoagulants
* Patients must not have any of following:

  * Cirrhosis at a level of Child-Pugh B (or worse);
  * Cirrhosis (any degree) and a history of hepatic encephalopathy; or
  * Clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Patients must have received exactly one line of anti-PD-1 or anti-PD-L1 therapy for at least 84 days as their most recent line of therapy, either alone or in combination with platinum-based chemotherapy. Patients must have experienced disease progression during or after this regimen. Patients whose most recent line of therapy was anti-PD-1 or anti-PD-L1 monotherapy must have also experienced disease progression during or after prior platinum-based chemotherapy
* Patients must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to substudy randomization. Patients must have recovered (=< grade 1) from any side effects of prior therapy, except for alopecia. Patients must not have received any radiation therapy within 14 days prior to sub-study randomization
* Patients must not have received nitrosoureas or mitomycin-c within 42 days prior to sub-study randomization
* Patients must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within seven days prior to sub-study randomization. Inhaled or topical steroids, and adrenal replacement doses =< 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Patients must not have received a live attenuated vaccination within 28 days prior to sub-study randomization
* Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Patients must not be receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents within 7 days prior to randomization. Once-daily aspirin use (maximum dose 325 mg/day) is permitted
* Patient must not have received radiotherapy within 14 days before the first dose of study treatment or received lung radiation therapy of > 30 Gy within 6 months before the first dose of study treatment

  * Note: Participants must have recovered from all radiation-related toxicities to grade 1 or less, not require corticosteroids, and not have had radiation pneumonitis
* Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to substudy randomization. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study randomization. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to sub-study randomization. CT and MRI scans must be submitted for central review via transfer of images and data (TRIAD)
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study randomization. Patient must not have leptomeningeal disease, spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to sub-study randomization, AND (2) patient has no residual neurological dysfunction and has been off corticosteroids for at least seven days prior to sub-study randomization
* Absolute neutrophil count (ANC) >= 1,500/mcl (obtained within 28 days prior to sub-study randomization)
* Platelet count >= 100,000 mcl (obtained within 28 days prior to sub-study randomization)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to sub-study randomization)
* Serum bilirubin =< institutional upper limit of normal (IULN) within 28 days prior to sub-study randomization. For patients with liver metastases, bilirubin must be =< 5 x IULN; and either
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN within 28 days prior to sub-study randomization (if both ALT and AST are done, both must be < 2 IULN). For patients with liver metastases, either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN)
* Serum creatinine =< the IULN OR calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to sub-study randomization
* Patients? urinary protein must be =< 1+ on dipstick or routine urinalysis (UA). If urine dipstick or routine analysis indicated proteinuria >= 2+, then a 24-hour urine is to be collected and demonstrate < 1000 mg of protein in 24 hours to allow participation in the study
* Patients must not have a history of uncontrolled or poorly-controlled hypertension (defined as >= 150 / >= 90 mm Hg for > 4 weeks) despite standard medical management
* International normalized ratio (INR) =< 1.5 (documented within 28 calendar days prior to randomization)
* Partial thromboplastin time (PTT) =< 5 seconds above the institutional upper limit of normal (IULN) (unless receiving anticoagulation therapy) (documented within 28 calendar days prior to randomization)
* Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile 14 days prior to randomization. If receiving warfarin, the patient must have an INR =< 3.0. For heparin and low molecular weight heparin (LMWH) there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices)
* Patients must have Zubrod performance status 0-1 documented within 28 days prior to sub-study randomization
* Pre-study history and physical exam must be obtained within 28 days prior to substudy randomization
* Patients must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method during the study and 4 months after study completion. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures during the study and 4 months after study completion
* Patients must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Patients must also be offered participation in banking and in the correlative studies for collection and future use of specimens
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Reckamp, Principal Investigator — SWOG Cancer Research Network
Locations (889):
- United States (889):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Loyola Center for Cancer Care and Research, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Saint Claire Regional Medical Center, Morehead, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 participants were initially randomized to the study, 82 to the ramucirumab + pembrolizumab (RP) arm and 84 to the standard of care (SOC) arm. 30 were ineligible, 13 in the RP arm and 17 in the SOC arm. In all, 136 participants were eligible and included in the primary analysis (RP n=69, SOC n=67).
Groups:
- Standard of Care (Inv. Choice): Participants receive investigator's choice of standard of care chemotherapy. Allowed regimens include docetaxel (75 mg/m2) IV; ramucirumab (10 mg/kg) plus docetaxel (75 mg/m2) IV once every 21 days; gemcitabine (1,000 mg/m2) IV on days 1 and 8 every 21 days; or for nonsquamous NSCLC patients only, pemetrexed (500 mg/m2) IV once every 21 days. Treatment continues until disease progression as defined in RECIST 1.1, symptomatic deterioration, unacceptable toxicity, treatment delay for any reason >84 days, or participant choice.
- Ramucirumab + Pembrolizumab: Participants receive open label ramucirumab (10 mg/kg intravenous [IV]) plus pembrolizumab (200 mg IV) once every 21 days. Treatment continues until disease progression as defined in RECIST 1.1, symptomatic deterioration, unacceptable toxicity, treatment delay for any reason >84 days, or participant choice.
Period: Overall Study
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Started | 67 | 69
Completed | 0 | 0
Not Completed | 67 | 69
Not completed — Adverse Event | 11 | 7
Not completed — Refusal unrelated to adverse event | 5 | 1
Not completed — Progression/relapse | 40 | 47
Not completed — Death | 6 | 3
Not completed — Other - not protocol specified | 5 | 4
Not completed — On treatment | 0 | 7

BASELINE CHARACTERISTICS:
Population: Participants who are eligible and evaluable for the primary analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Median (Full Range); unit: years] | 65.8 [45.6 to 84.3] | 66.4 [37.6 to 85.3] | 65.9 [37.6 to 85.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 42 | 41 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 66 | 66 | 132
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 58 | 60 | 118
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 18 | 19 | 37
  Past Smoker | 43 | 44 | 87
  Never Smoked | 6 | 6 | 12
Performance Status [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status scale:
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 9 | 23 | 32
    1 | 58 | 46 | 104
Tumor Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 39 | 36 | 75
  Squamous cell | 27 | 28 | 55
  Mixed < 50% squamous cell | 1 | 0 | 1
  Mixed >= 50% squamous cell | 0 | 1 | 1
  Other non-small-cell, NOS | 0 | 4 | 4
Prior Lines of Treatment for Stage IV Disease [Count of Participants; unit: Participants]
  0 | 4 | 4 | 8
  1 | 33 | 35 | 68
  2 | 17 | 19 | 36
  >= 3 | 13 | 11 | 24
PD-L1 Status [Count of Participants; unit: Participants] — Population: Percentages are calculated among those with known status only. 10 participants had unknown PD-L1 status.
  Participants
    number analyzed (Participants) | 64 | 62 | 126
    < 1% | 26 | 29 | 55
    1% - 49% | 22 | 21 | 43
    >= 50% | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time from date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: From date of registration to a maximum of 2 years and 11 months or death
Population: Eligible and evaluable participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
months | 11.6 [9.9 to 13.0] | 14.5 [13.9 to 16.1]
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Comparison of OS was performed using a standard stratified log-rank test and a weighted log-rank test. The study had 90% power to detect the scenario with overlapping curves up to 3 months and a hazard ratio of 0.5 after 3 months, assuming exponentially distributed survival times, a median OS of 10.5 months in the SOC arm, and uniform accrual over 21-24 months. This analysis reports the standard stratified log-rank test; Test type: Superiority; p = 0.05, Log Rank — If either P value from the two tests (standard stratified log-rank and weighted log-rank) was < 0.0972, the study would be considered to have rejected the null at the one-sided 10% level; Testing was performed using a standard stratified log-rank test; Hazard Ratio (HR) = 0.69, 80% CI 2-sided [0.51 to 0.92] — Treatment effects comparing the RP arm to the SOC arm were summarized using a Cox proportional hazards model including the stratification factors (PD-L1 status and histology) and 80% CIs
Statistical Analysis 2: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Comparison of OS was performed using a standard stratified log-rank test and a weighted log-rank test. The study had 90% power to detect the scenario with overlapping curves up to 3 months and a hazard ratio of 0.5 after 3 months, assuming exponentially distributed survival times, a median OS of 10.5 months in the SOC arm, and uniform accrual over 21-24 months. This analysis reports the weighted log-rank test; Test type: Superiority; p = 0.15, Log Rank — If either p-value from the two tests (standard stratified log-rank and weighted log-rank) was < 0.0972, the study would be considered to have rejected the null at the one-sided 10% level

2. Secondary Outcome: Response Rate (RR)
Description: Percentage of participants with a complete or partial, confirmed or unconfirmed response.
  Complete Response (CR): Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  Partial Response (PR): Applies only to participants with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
Percentage of participants | 28 [19 to 37] | 22 [14 to 30]
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Test type: Superiority; p = 0.19, Chi-squared — Proportions were compared using a chi-squared test at the one-sided 5% level

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with complete response (CR), partial response (PR), or stable disease as best response.
  CR: Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes must have reduction in short axis to <1.0cm. All disease must be assessed using the same technique as baseline.
  PR: Applies only to participants with at least one measurable lesion. At least 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
  Stable disease: Does not qualify for CR, PR, Progression or Symptomatic Deterioration. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
Percentage of participants | 73 [64 to 82] | 75 [67 to 84]
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Test type: Superiority; p = 0.38, Chi-squared — Proportions were compared using a chi-squared test at the one-sided 5% level

4. Secondary Outcome: Duration of Response (DOR)
Description: Time from date of first documentation of response (complete or partial) to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause among participants who achieve a response. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan (as defined by the disease assessment schedule) is used as the date of progression.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants who had a response
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 19 | 15
months | 5.6 [4.6 to 7.8] | 12.9 [2.8 to NA] — Insufficient number of participants with events

5. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drugs are reported. CTCAE Version 5.0 was used for all AE reporting.
Time Frame: Duration of treatment and follow-up until death or 3 years post randomization
Population: Participants who were eligible and received at least one dose of protocol treatment
Measure: Number; unit: Participants
Groups:
- Standard of Care (Inv. Choice): Participants receive investigatorXXs choice of standard of care chemotherapy. Allowed regimens include docetaxel (75 mg/m2) IVXX ramucirumab (10 mg/kg) plus docetaxel (75 mg/m2) IV once every 21 daysXX gemcitabine (1,000 mg/m2) IV on days 1 and 8 every 21 daysXX or for nonsquamous NSCLC patients only, pemetrexed (500 mg/m2) IV once every 21 days. Treatment continues until disease progression as defined in RECIST 1.1, symptomatic deterioration, unacceptable toxicity, treatment delay for any reason >84 days, or participant choice.
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 60 | 69
Participants
  Abdominal infection | 1 | 0
  Acidosis | 1 | 0
  Acute kidney injury | 1 | 4
  Adrenal insufficiency | 0 | 2
  Alanine aminotransferase increased | 2 | 1
  Anemia | 4 | 0
  Anorexia | 1 | 0
  Arterial thromboembolism | 0 | 1
  Arthralgia | 0 | 2
  Ascites | 1 | 1
  Aspartate aminotransferase increased | 2 | 2
  Blood bilirubin increased | 0 | 2
  Bronchopulmonary hemorrhage | 0 | 1
  Cardiac arrest | 0 | 1
  Colitis | 1 | 0
  Colonic perforation | 2 | 0
  Cough | 0 | 1
  Creatinine increased | 0 | 1
  Death NOS | 0 | 1
  Dehydration | 3 | 0
  Delirium | 0 | 1
  Diarrhea | 2 | 0
  Dizziness | 1 | 0
  Duodenal ulcer | 1 | 0
  Dyspnea | 3 | 3
  Encephalopathy | 0 | 1
  Fatigue | 4 | 4
  Febrile neutropenia | 3 | 1
  Gastric hemorrhage | 1 | 1
  Gastrointestinal disorders - Other, specify | 1 | 0
  Generalized muscle weakness | 0 | 2
  Hypertension | 2 | 9
  Hypoalbuminemia | 2 | 0
  Hypokalemia | 1 | 1
  Hypomagnesemia | 0 | 1
  Hyponatremia | 0 | 1
  Hypophosphatemia | 1 | 0
  Hypotension | 3 | 0
  Hypoxia | 2 | 2
  Infusion related reaction | 0 | 1
  Lung infection | 4 | 4
  Lymphocyte count decreased | 11 | 3
  Mucositis oral | 4 | 0
  Multi-organ failure | 1 | 0
  Muscle weakness lower limb | 1 | 0
  Nausea | 3 | 1
  Neutrophil count decreased | 20 | 3
  Pericardial effusion | 1 | 0
  Peripheral sensory neuropathy | 0 | 1
  Platelet count decreased | 3 | 0
  Pleural effusion | 1 | 0
  Pneumonitis | 1 | 1
  Pneumothorax | 0 | 1
  Portal hypertension | 1 | 0
  Proteinuria | 0 | 2
  Respiratory failure | 2 | 2
  Sepsis | 5 | 3
  Sinus tachycardia | 0 | 1
  Stroke | 1 | 0
  Syncope | 0 | 1
  Thromboembolic event | 2 | 1
  Vomiting | 2 | 0
  Weight loss | 0 | 1
  Wheezing | 0 | 2
  White blood cell decreased | 17 | 1

6. Secondary Outcome: Investigator Assessed-progression-free Survival (IA-PFS)
Description: Time from date of registration to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan is used as the date of progression.
  Symptomatic deterioration: Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression. Efforts should be made to obtain objective evidence of progression after discontinuation.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
months | 5.2 [4.2 to 5.7] | 4.5 [4.2 to 6.1]
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Comparison of IA-PFS was performed using a standard stratified log-rank test and a weighted log-rank test with weights equal to 1-S(t), where S(t) is the pooled survival estimate at time t (G[rho=0, gamma=1]). The weighted test weights later events over earlier events and has more power than the standard log-rank test under a delayed separation in the curves. This analysis reports the standard stratified log-rank test; Test type: Superiority; p = 0.25, Log Rank; Testing was performed using a standard stratified log-rank test; Hazard Ratio (HR) = 0.86, 80% CI 2-sided [0.66 to 1.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; Comparison of IA-PFS between the RP and SOC arms was performed using a standard stratified log-rank test and a weighted log-rank test with weights equal to 1-S(t), where S(t) is the pooled survival estimate at time t (G[rho=0, gamma=1]). The weighted test weights later events over earlier events and has more power than the standard log-rank test under a delayed separation in the curves. This analysis reports the weighted log-rank test; Test type: Superiority; p = 0.14, Log Rank; Testing was performed using a weighted log-rank test

7. Secondary Outcome: Overall Survival (OS), Subgroup Analysis by Stratification Factors
Description: Number of participants who died due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number; unit: Participants
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
Participants
  PD-L1: < 1%: number analyzed (Participants) | 26 | 29
  PD-L1: < 1% | 21 | 21
  PD-L1: >= 1%: number analyzed (Participants) | 38 | 33
  PD-L1: >= 1% | 27 | 19
  Histology: Squamous: number analyzed (Participants) | 28 | 29
  Histology: Squamous | 24 | 18
  Histology: Non-squamous: number analyzed (Participants) | 39 | 40
  Histology: Non-squamous | 27 | 27
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the PD-L1 < 1% subgroup; Test type: Superiority; p = 0.16, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.74, 80% CI 2-sided [0.50 to 1.10] — Treatment effects comparing the RP arm to the SOC arm were summarized using a Cox proportional hazards model and 80% CIs
Statistical Analysis 2: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the PD-L1 >= 1% subgroup; Test type: Superiority; p = 0.08, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.66, 80% CI 2-sided [0.45 to 0.97] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the squamous histology subgroup; Test type: Superiority; p = 0.005, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.43, 80% CI 2-sided [0.28 to 0.65] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the non-squamous histology subgroup; Test type: Superiority; p = 0.43, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.95, 80% CI 2-sided [0.67 to 1.35] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Investigator-Assessed Progression-Free Survival (IA-PFS), Subgroup Analysis by Stratification Factors
Description: Number of participants with progression assessed by local review or symptomatic deterioration, or death due to any cause. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan is used as the date of progression.
  Symptomatic deterioration: Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression. Efforts should be made to obtain objective evidence of progression after discontinuation.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number; unit: Participants
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 67 | 69
Participants
  Histology: Non-squamous: number analyzed (Participants) | 39 | 40
  Histology: Non-squamous | 34 | 34
  Histology: Squamous: number analyzed (Participants) | 28 | 29
  Histology: Squamous | 28 | 23
  PD-L1: < 1%: number analyzed (Participants) | 26 | 29
  PD-L1: < 1% | 25 | 27
  PD-L1: >= 1%: number analyzed (Participants) | 38 | 33
  PD-L1: >= 1% | 34 | 24
Statistical Analysis 1: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the PD-L1 < 1% subgroup; Test type: Superiority; p = 0.28, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.84, 80% CI 2-sided [0.58 to 1.22] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the PD-L1 >= 1% subgroup; Test type: Superiority; p = 0.07, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.67, 80% CI 2-sided [0.48 to 0.95] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the squamous histology subgroup; Test type: Superiority; p = 0.02, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.55, 80% CI 2-sided [0.38 to 0.80] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Standard of Care (Inv. Choice) vs Ramucirumab + Pembrolizumab; This analysis includes the results for the non-squamous histology subgroup; Test type: Superiority; p = 0.41, Log Rank — One-sided p-values were calculated using a standard log-rank test; Hazard Ratio (HR) = 0.95, 80% CI 2-sided [0.69 to 1.29] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 3 years post randomization, whichever occurs first.
Description: CTCAE Version 5.0 was used for routine toxicity reporting and Serious Adverse Event (SAE) reporting. 129 participants were treated and evaluated for AEs: 69 on the Ramucirumab + Pembrolizumab arm and 60 on the Standard of Care arm.
  All-cause mortality is reported for all eligible participants (69 on the Ramucirumab + Pembrolizumab arm and 67 on the Standard of Care arm), including those who did not receive protocol treatment.
Arm/Group | Standard of Care (Inv. Choice) | Ramucirumab + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 51/67 | 45/69
Serious Adverse Events (participants affected / at risk) | 11/60 | 28/69
Other Adverse Events (participants affected / at risk) | 60/60 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (Inv. Choice) (N=60) | Ramucirumab + Pembrolizumab (N=69)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Death NOS (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Fever (General disorders) | 0 | 2
Infusion site extravasation (General disorders) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 7
Sepsis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Cardiac troponin I increased (Investigations) | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Weight loss (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Neoplasms benign, malignant and unspecified (incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial thromboembolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 5
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (Inv. Choice) (N=60) | Ramucirumab + Pembrolizumab (N=69)
Anemia (Blood and lymphatic system disorders) | 40 | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Sinus tachycardia (Cardiac disorders) | 9 | 5
Hypothyroidism (Endocrine disorders) | 1 | 18
Dry eye (Eye disorders) | 4 | 1
Watering eyes (Eye disorders) | 16 | 2
Abdominal pain (Gastrointestinal disorders) | 15 | 8
Ascites (Gastrointestinal disorders) | 3 | 2
Colonic perforation (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 12 | 12
Diarrhea (Gastrointestinal disorders) | 29 | 19
Dry mouth (Gastrointestinal disorders) | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 2
Mucositis oral (Gastrointestinal disorders) | 19 | 3
Nausea (Gastrointestinal disorders) | 24 | 23
Oral pain (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 14 | 13
Chills (General disorders) | 8 | 5
Edema limbs (General disorders) | 14 | 9
Fatigue (General disorders) | 42 | 39
Fever (General disorders) | 10 | 6
Flu like symptoms (General disorders) | 3 | 2
Non-cardiac chest pain (General disorders) | 5 | 2
Pain (General disorders) | 8 | 10
Infections and infestations-Other (Infections and infestations) | 3 | 8
Lung infection (Infections and infestations) | 10 | 5
Sepsis (Infections and infestations) | 5 | 0
Sinusitis (Infections and infestations) | 4 | 1
Skin infection (Infections and infestations) | 3 | 5
Thrush (Infections and infestations) | 5 | 0
Upper respiratory infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Bruising (Injury, poisoning and procedural complications) | 5 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 9 | 6
Alkaline phosphatase increased (Investigations) | 13 | 14
Aspartate aminotransferase increased (Investigations) | 11 | 9
Blood bilirubin increased (Investigations) | 5 | 4
Creatinine increased (Investigations) | 11 | 11
Investigations-Other (Investigations) | 10 | 5
Lymphocyte count decreased (Investigations) | 24 | 13
Neutrophil count decreased (Investigations) | 26 | 6
Platelet count decreased (Investigations) | 17 | 19
Thyroid stimulating hormone increased (Investigations) | 2 | 10
Weight loss (Investigations) | 15 | 17
White blood cell decreased (Investigations) | 27 | 11
Anorexia (Metabolism and nutrition disorders) | 22 | 24
Dehydration (Metabolism and nutrition disorders) | 7 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 11 | 6
Hypernatremia (Metabolism and nutrition disorders) | 2 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 | 31
Hypocalcemia (Metabolism and nutrition disorders) | 11 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalemia (Metabolism and nutrition disorders) | 11 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatremia (Metabolism and nutrition disorders) | 17 | 27
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Dizziness (Nervous system disorders) | 15 | 13
Dysgeusia (Nervous system disorders) | 13 | 7
Headache (Nervous system disorders) | 15 | 16
Lethargy (Nervous system disorders) | 2 | 4
Paresthesia (Nervous system disorders) | 5 | 2
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 5
Anxiety (Psychiatric disorders) | 6 | 2
Confusion (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 10 | 5
Hematuria (Renal and urinary disorders) | 3 | 7
Proteinuria (Renal and urinary disorders) | 14 | 27
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 8
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6
Nail changes (Skin and subcutaneous tissue disorders) | 6 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 7
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 9 | 3
Hypertension (Vascular disorders) | 15 | 23
Hypotension (Vascular disorders) | 8 | 8
Thromboembolic event (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03971474/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03971474/ICF_001.pdf